CLINICAL TRIAL: NCT01368718
Title: The Effect of Nasal CPAP in Patients With Chronic Fatigue and Sleep-disordered Breathing
Brief Title: Nasal Continuous Positive Airway Pressure (CPAP) in Chronic Fatigue and Sleep-disordered Breathing
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low inclusion and adherence rates
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2011/191
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Chronic Fatigue With OSA; Chronic Fatigue Syndrome With OSA

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active/Sham CPAP (Other)
  Interventions: Procedure: Active CPAP is compared with sham CPAP as a control intervention.

INTERVENTIONS:
Procedure: Active CPAP is compared with sham CPAP as a control intervention. — Patients are randomized into active or control arm. After the first treatment, a washout period is installed,after which therapy is switched according to the cross-over protocol. A CPAP device consists of a unit that generates airflow, which is directed to the airway via a mask. With active CPAP, the generated airflow creates a positive pressure and prevents upper airway collapse. With sham CPAP, the generated airflow creates a very low pressure.

SUMMARY:
Chronic fatigue (CF) and chronic fatigue syndrome (CFS) are disabling disorders that may be induced or aggravated by underlying sleep disturbances. The relationship between sleep quality and fatigue is still not fully elucidated. To evaluate the effect of improved sleep quality on fatigue, a randomized controlled and cross-over trial with nasal continuous positive airway pressure (nCPAP) is carried out in patients who present with a primary complaint of chronic disabling fatigue and who are found to have an apnea-hypopnea index (AHI) >= 15 on polysomnography (PSG).

The aim of this study is to address the issue of Continuous Positive Airway Pressure-responsiveness regarding fatigue as a presenting symptom in CF and CFS patient with obstructive sleep apnea (OSA), in the absence of underlying medical or psychiatric illness. The answer to this question may shed further light on the enigmatic relationship between sleep and fatigue. We also want to investigate the Continuous Positive Airway Pressure responsiveness regarding sleepiness and general health in the same target population. Zero-hypothesis: there is no effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients primarily referred for disabling, unexpected fatigue.
* According to the Fukuda criteria, diagnostic work-up yields a final diagnosis of chronic fatigue (CF) or chronic fatigue syndrome (CFS).
* 18 <= age <= 65
* Polysomnography Test (PSG) demonstrates an apnea-hypopnea index (AHI) >=15, as evidence for obstructive sleep apnea (OSA).
* Female patient of childbearing potential (premenopausal female biologically capable of becoming pregnant) has a confirmed negative pregnancy test at the start of the Continuous Positive Airway Pressure (CPAP) trial and has to employ an acceptable method of birth control.
* Written, signed and dated informed consent must be obtained from each patient.
* Patient able to understand and follow the requirements of the study and to comply.
* Willing to abstain from taking any medication or treatment prohibited in the protocol.

Exclusion Criteria:

* Patients primarily referred for Excessive Daytime Sleepiness (EDS) or snoring.
* Fatigue that is explained by medical or psychiatric causes.
* 18 > age > 65
* Apnea-Hypopnea Index (AHI) < 15
* Body Mass Index (BMI) >= 40, calculated as weight(m)/(height (m))²
* Parasomnia
* Severe sleepiness with (Epworth Sleepiness Scale) ESS >= 16 (=15% of the Chronic fatigue syndrome (CFS) population)
* Tonsillar hypertrophy (Friedman grade III and IV tonsils)
* Signs of nasal obstruction, including chronic use of topical nasal drugs.
* Earlier CPAP treatment
* Physical and mental disability that compromises the normal use of CPAP
* CPAP intolerance
* Current use of sedative (benzodiazepine and non-benzodiazepine GABA-esgic agonist) or antidepressant medication for a time period inferior to 3 weeks.
* Female patient who is pregnant, lactating or has a positive pregnancy test result.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2017-04-11 (Actual)

PRIMARY OUTCOMES:
Continuous Positive Airway Pressure-responsiveness regarding fatigue after 28 days: baseline evaluation. | At day 0
  Baseline evaluation before treatment. Questionnaires Fatigue Severity Scale (FSS), Checklist Individual Strength(CIS), Visual Analogue Scale for Fatigue (VAS-F) are used.
Continuous Positive Airway Pressure-responsiveness regarding fatigue after 28 days: first treatment + effect evaluation. | Treatment takes 28 days after first evaluation
  At the end of the first treatment: effect evaluation. Questionnaires Fatigue Severity Scale (FSS), Checklist Individual Strength(CIS), Visual Analogue Scale for Fatigue (VAS-F) are used.
Continuous Positive Airway Pressure-responsiveness regarding fatigue after 28 days: second treatment + effect evaluation. | Treatment takes 28 days after second evaluation
  At the end of the second treatment: effect evaluation. Questionnaires Fatigue Severity Scale (FSS), Checklist Individual Strength(CIS), Visual Analogue Scale for Fatigue (VAS-F) are used.

SECONDARY OUTCOMES:
The Continuous Positive Airway Pressure responsiveness regarding sleepiness and general health in the same target population: baseline evaluation. | At day 0
  Before treatment: baseline evaluation. Polysomnography Test (PSG) , Multiple Sleep Latency Test (MSLT) and questionnaires ( Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), Medical Outcomes Study Short Form 36-item (MOS SF36)) are used.
The Continuous Positive Airway Pressure responsiveness regarding sleepiness and general health in the same target population: first treatment + effect evaluation. | Treatment takes 28 days after first evaluation
  At the end of the first treatment: effect evaluation. Polysomnography Test (PSG) , Multiple Sleep Latency Test (MSLT) and questionnaires ( Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), Medical Outcomes Study Short Form 36-item (MOS SF36)) are used.
The Continuous Positive Airway Pressure responsiveness regarding sleepiness and general health in the same target population: second treatment + effect evaluation. | Treatment takes 28 days after second evaluation
  At the end of the second treatment: effect evaluation. Polysomnography Test (PSG) , Multiple Sleep Latency Test (MSLT) and questionnaires ( Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), Medical Outcomes Study Short Form 36-item (MOS SF36)) are used.

CONTACTS AND LOCATIONS:
Overall Officials: An Mariman, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium